CLINICAL TRIAL: NCT02664870
Title: Prospective Biological and Clinical Databank for the Evaluation of Biomarkers in Human Synovial Fluid
Brief Title: Evaluation of Biomarkers in Human Synovial Fluid
Status: Active, not recruiting | Type: Observational
Sponsor: Duke University (Other)
Responsible Party: Sponsor
Other Study IDs: Pro00066468
Record Dates: First submitted 2016-01-07; First posted 2016-01-27 (Estimated); Last update posted 2026-02-04 (Actual); Status verified 2026-02

CONDITIONS: Osteoarthritis
Keywords: synovial fluid; biomarkers
MeSH Terms: conditions — Osteoarthritis | interventions — Arthroscopy; Arthroplasty

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Biospecimen retention would include the collection and storage of synovial fluid samples from the hip, shoulder, and knee.
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- Shoulder Patients: Patients (1) without evidence of cartilage damage, (2) with molecular change, (3) physiologic change, or (4) with end-stage osteoarthritis, who require arthroscopy or arthroplasty
  Interventions: Procedure: Arthroscopy; Procedure: Arthroplasty
- Hip Patients: Patients (1) without evidence of cartilage damage, (2) with molecular change, (3) physiologic change, or (4) with end-stage osteoarthritis, who require arthroscopy (with or without periacetabular osteotomy (PAO)) or arthroplasty
  Interventions: Procedure: Arthroscopy; Procedure: Arthroplasty
- Knee Patients: Patients (1) without evidence of cartilage damage, (2) with molecular change, (3) physiologic change, or (4) with end-stage osteoarthritis, who require arthroscopy or arthroplasty
  Interventions: Procedure: Arthroscopy; Procedure: Arthroplasty

INTERVENTIONS:
Procedure: Arthroscopy — Arthroscopic Surgery on the hip, shoulder, or knee
Procedure: Arthroplasty — Total hip, shoulder, or knee arthroplasty

SUMMARY:
Osteoarthritis is a condition that causes joints in the human body to deteriorate over time. This condition affects more than 250 million people around the globe. Currently, the goal of treating osteoarthritis involves reducing the severity and pain that results from the disease. The ultimate goal of this study is to identify patients with pre-arthritic joints (before symptoms or disease characteristics appear) in an effort to find and use treatments that stop or slow the disease. Joints are filled with a naturally occurring liquid known as synovial fluid. Molecules (biomarkers) and genetic expression of various cell types within synovial joint fluid may serve as measures of onset and progression of osteoarthritis. These samples have the potential to improve diagnosis, classification, and treatment, possibly changing the natural history of this debilitating disease. The purpose of this study is to develop a collection of synovial fluid samples from the shoulder, hip and knee for the analysis of biomarkers and cellular and genetic components therein to better understand the pre-arthritic joint, progression to disease, and response to interventions.

ELIGIBILITY:
Inclusion Criteria:

1. Adult patients ( > 18 years old)
2. Patient is eligible for general anesthesia and either arthroscopy or arthroplasty.
3. Patient needs standard of care arthroscopy or arthroplasty of either shoulder, hip or knee joint for osteoarthritis or prearthritic conditions.
4. Patient must have signed an IRB approved informed consent document for the arthrocentesis procedure which will be performed during the arthroscopic or arthroplastic procedure.

Exclusion Criteria:

1. Active Joint Infection within last 6 months.
2. Previous arthroplasty in the joint undergoing arthroplasty
3. History of auto-immune arthropathies.
4. History of HIV or Hepatitis C

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients will be recruited at the Sports Medicine and Adult Reconstruction Clinics at Duke University Medical Center.
Sampling Method: Non-Probability Sample
Enrollment: 149 (Actual)
Dates: Start 2016-01; Primary Completion 2019-01-24 (Actual); Study Completion 2028-01-01 (Estimated)

PRIMARY OUTCOMES:
Feasibility of biobank data collection as measured by percentage of patients with a complete data set one year post-operation | 1 year
  Study participants will be enrolled over an anticipated time frame of 2 years. One year following the last participant's enrollment prompts an anticipated three year time frame to determine the feasibility of biobank data collection.

SECONDARY OUTCOMES:
Number of biomarkers worthy of study to aid in the diagnosis and progression of osteoarthritis | 3-5 years
  Biomarkers for study include the following: CRP, Eotaxin, Eotaxin-3, FGF (basic), Flt-1/VEGFR1, GM-CSF, ICAM-1, IFN-γ, IL-10, IL-12/IL-23p40, IL-12p70, IL-13, IL-15, IL-16, IL-17A, IL-1α, IL-1β, IL-2, IL-4, IL-5, IL-6, IL-7, IL-8, IL-8 (HA), IP-10, MCP-1, MCP-4, MDC, MIP-1α, MIP-1β, PlGF, SAA, TARC, Tie-2, TNF-α, TNF-β, VCAM-1, VEGF-A, VEGF-C, VEGF-D, clusterin, lubricin, and matrix molecules.
Types of biomarkers worthy of study to aid in the diagnosis and progression of osteoarthritis | 3-5 years
  Types of biomarkers include the following: chemokines, cytokines, inflammatory, angiogenesis, and vascular injury.
Number of patients who responded to non-arthroplasty intervention based on biomarker analysis and measured with questionnaires | 1-10 years
Number of patients who did not respond to non-arthroplasty intervention based on biomarker analysis and measured with questionnaires | 1-10 years

CONTACTS AND LOCATIONS:
Overall Officials: Richard C. Mather, MD, MBA, Principal Investigator — Duke University
Locations (1):
- Duke Orthopaedic Clinics, Durham, North Carolina, United States